CLINICAL TRIAL: NCT05313152
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAVO103A in Adult Healthy Subjects
Brief Title: Study of TAVO103A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tavotek Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 59870002
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TAVO103A Low Dose (Experimental): TAVO103A: TAVO103A single ascending dose IV infusion.
  Interventions: Drug: TAVO103A
- TAVO10A Medium Dose (Experimental): TAVO103A: TAVO103A single ascending dose IV infusion.
  Interventions: Drug: TAVO103A
- TAVO103A High Dose (Experimental): TAVO103A: TAVO103A single ascending dose IV infusion.
  Interventions: Drug: TAVO103A
- Placebo (Placebo Comparator): Placebo single ascending dose IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TAVO103A — TAVO103A single ascending dose IV infusion.
  Arms: TAVO103A High Dose; TAVO103A Low Dose; TAVO10A Medium Dose
Other: Placebo — Placebo single ascending dose IV infusion.
  Arms: Placebo

SUMMARY:
This is a Phase 1, single ascending dose study designed to investigate TAVO103A, administered as an IV infusion up to 60 minutes in length to healthy adult subjects. This study is designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TAVO103A.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD), single site study. There will be up to 5 SAD cohorts with 6 subjects enrolled into each. Subjects will be randomized at a ratio of 2:1 to receive TAVO103A or placebo. Subjects will be evaluated for safety throughout the study up through day 196.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 and ≤ 65 years of age, inclusive.
* Subjects must have a body weight range of ≥ 50 kg and ≤ 100 kg, inclusive, and a BMI ≥ 18.0 and ≤ 30.0 kg/m2, inclusive.
* Subjects must be healthy based on clinical laboratory tests performed at Screening and Day -1.
* Females of childbearing potential who are sexually active with a male partner must agree to use a highly effective method of contraception from screening through the end of the study.
* Males who are sexually active and nonsterile, and whose partners are females of childbearing potential must agree to use condoms from screening through the end of the study.
* Males must agree to not donate sperm from screening through the end of the study.
* Subjects must be able to communicate effectively with the study personnel.
* Subjects must be nonsmokers, defined as having abstained from tobacco- or nicotine-containing products in the 6 months prior to Screening.
* Subjects will be considered eligible according to the following tuberculosis screening criteria's.
* Subjects must sign an informed consent form.

Exclusion Criteria:

* Positive pregnancy test or is lactating at any time during the study.
* History or presence of conditions which, in the judgment of the investigator, are known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History or presence of conditions that may place the subject at increased risk as determined by the investigator.
* Subject currently has or has had a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the subject.
* Subject has a QT corrected according to Fridericia's formula (QTcF) interval > 450 msec (males) or > 470 msec (for females), has a complete left or right bundle branch block, or has a history or current evidence of additional risk factors for Torsades de Pointes.
* History of surgery or major trauma within 16 weeks of Screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study, or within 17 weeks after the last dose of study drug administration.
* Subject plans to undergo non-major elective surgery within 4 weeks prior to study drug administration through EOS.
* Subject has a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies or antibody fragments, or to any components of the formulation of TAVO103A and its excipients used in this study.
* History of alcohol abuse, illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of Screening.
* Use of prescription medications within 14 days or any drugs that induce or inhibit study drug-specific cytochrome 450(s) within 14 days or 5 half-lives (if known), whichever is longer, prior to administration of the study drug. By exception, prescription drugs, such as hormonal birth control or hormone replacement therapy, will be permitted.
* Use of OTC drugs (including herbal preparations) within 7 days or 5 half-lives (if known), whichever is longer, prior to administration of the study drug. Common OTC drugs are acceptable with investigator approval.
* Has received a vaccination within 30 days prior to administration of the study drug
* Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug's PK, PD, or biological activity (if known), whichever is longer, prior to administration of the study drug in this study or is currently participating in another clinical study.
* Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
* Strenuous activity within 48 hours prior to CRU admission.
* Consumption of alcohol or caffeine-containing food or beverages within 3 days prior to CRU admission
* Positive urine drugs of abuse, alcohol breath test, or cotinine screen at any time during the study.
* Positive test for HIV-1 or HIV-2 antibodies.
* Positive test for hepatitis B virus or hepatitis C virus consistent with current infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
The severity of adverse effects according to the CTCAE Guidance for Industry, Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO103A in healthy volunteers. The Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials will be graded according to the National Cancer Institute's Common Terminology Criteria for AEs, Version 5.0. Which will have a minimum value of Grade 1, or mild, and a maximum value of Grade 4, or Potentially Life Threatening.
Changes in vital signs including oral temperature or tympanic temperature (C°) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO103A in healthy volunteers.
Changes in vital signs including respiratory rate (breaths per minute) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO103A in healthy volunteers.
Changes in vital signs including systolic and diastolic blood pressure (mmHg) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO103A in healthy volunteers.
Changes in vital signs including pulse rate (beats per minute) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO103A in healthy volunteers.

SECONDARY OUTCOMES:
Immunogenicity of TAVO103A [Time Frame: Day 1 through Day 196] | 196 days
  Incidence of anti-drug antibodies (ADA) following dosing of TAVO103A
Cmax (Maximum observed serum concentration ) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
tmax (time that Cmax was observed) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
AUC-last (Area under the serum concentration-time curve from time 0 to the time of the last quantifiable concentration; calculated using the linear/log trapezoid rule) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
AUC-inf (Area under the serum concentration-time curve from time 0 extrapolated to infinity) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
AUC0-t (Area under the serum concentration-time curve from time 0 to time t) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
t½ (Terminal elimination half-life) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
λz (Terminal elimination rate constant) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
CL (Systemic clearance) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.
Vd (Volume of distribution) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the pharmacokinetics of TAVO103A in healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No